Document Date: 02-23-18

ID: H-41207

Title: A Window of Opportunity Trial: Avelumab in Non-metastatic Muscle Invasive

**Bladder Cancer** 

NCT03498196

## Statistical analysis

To see the change in T cells pre- and post-treatment, paired t-test or nonparametric Wilcoxon signed rank test will be used after checking its normality. Pathological response rate will be estimated along with 95% confidence interval. Two year disease free survival will be calculated using Kaplan-Meier survival curves with estimates of median and 95% confidence interval. Patients who are decided not to be evaluable for the primary outcome will be considered evaluable for the safety analysis and secondary outcomes, such patients will be summarized descriptively. The correlation of translational studies with response parameters will be summarized descriptively. Changes from pre- and post- treatment will be assessed using paired tests. SAS software will be used for all statistical analyses.